CLINICAL TRIAL: NCT01933035
Title: Extended Platelet Parameters as a Means to Differentiate Immune Thrombocytopenia From Hypo-proliferative Thrombocytopenias.
Status: Completed | Type: Observational
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-0134
Record Dates: First submitted 2013-08-28; First posted 2013-08-30 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Immune Thrombocytopenia; Chemotherapy Induced Thrombocytopenia; Myelodysplasia; Aplastic Anaemia
Keywords: ITP; Thrombocytopenia; mean platelet mass; mean platelet component
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Anemia, Refractory, with Excess of Blasts; Anemia, Aplastic; Thrombocytopenia | interventions — 1-methyl-1-piperidinomethane sulfonate; Population Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Study subjects will have the following collected: Lavender tri-potassium EDTA tubes filled according to the manufacturer's specifications [approximately 4ML of venous blood], labeled, and promptly dispatched to the laboratory.The sample will be gently inverted several times prior to analysis on the ADVIA 120 taking care not to overly agitate the sample. Moreover, the specimen shall be inspected for clot formation prior to being assayed. The full blood count shall be obtained and in the configuration sub-menu the extended platelet parameter option shall be selected and thus actuated. A print out will be generated including the MPC, MPM, platelet component distribution width, platelet mass distribution width, and large platelet count in addition to the standard platelet count and mean platelet volume [MPV].
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Immune Thrombocytopenics: The study shall be a single institution prospective cohort study. Comparison will be made among individuals with known ITP . Those with known hypo-proliferative forms of thrombocytopenia [aplastic anaemia, chemotherapy induced thrombocytopenia, and myelodysplastic thrombocytopenia, and a control population.
  Interventions: Other: Immune Thrombocytopenics
- Hypo-proliferative thrombocytopenics: The study shall be a single institution prospective cohort study. Comparison will be made between individuals with known ITP versus those with known hypo-proliferative forms of thrombocytopenia [aplastic anaemia, chemotherapy--induced thrombocytopenia, and myelodysplastic thrombocytopenia], and a control population.
  Interventions: Other: Hypo-proliferative thrombocytopenics
- Control Pupulation: comprised of healthy individuals with normal platelet counts, to confirm normal values for MPC and MPM
  Interventions: Other: Control Population

INTERVENTIONS:
Other: Immune Thrombocytopenics — Full blood count with extended platelet parameters
  Other Names: MPC (g/dl); MPM (pg)
  Groups: Immune Thrombocytopenics
Other: Hypo-proliferative thrombocytopenics — Full blood count with extended platelet parameters
  Other Names: MPC (g/dl); MPM (pg)
  Groups: Hypo-proliferative thrombocytopenics
Other: Control Population — Full blood count with extended platelet parameters
  Other Names: MPC (g/dl); MPM (pg)
  Groups: Control Pupulation

SUMMARY:
To utilise extended platelet parameters in order to individuate Immune Thrombocytopenia (ITP) from hypo-proliferative causes of thrombocytopenia.

To develop the clinical potential of the extended platelet parameters as they pertain to distinguishing different causes of thrombocytopenia from one another.

To test the hypothesis that mean platelet component (MPC) and mean platelet mass (MPM) might distinguish between thrombocytopenia related to bone marrow dysfunction and immune mediated destruction of platelets.

DETAILED DESCRIPTION:
Patient to be registered at the Haematology-Oncology department Mount Sinai Roosevelt Hospital.

Inclusion criteria are as follows:

All individuals age 18yrs and above capable of rendering consent Known ITP confirmed by response to IVIG, glucocorticoids, or WinRho and exclusion of all other possible causes of thrombocytopenia Confirmed aplastic anemia [as assessed through bone marrow trephine biopsy]. Chemotherapy-induced thrombocytopenia assessed at time of predicted nadir.

ELIGIBILITY:
Inclusion Criteria:

* All individuals age 18yrs and above capable of rendering consent
* Known ITP confirmed by response to intravenous immune globulin (IVIG), glucocorticoids, or winRho and exclusion of all other possible causes of thrombocytopenia
* Confirmed aplastic anemia [as assessed through bone marrow trephine biopsy]
* Chemotherapy induced thrombocytopenia assessed at time of predicted nadir.

Exclusion Criteria:

* Suspected multifactorial thrombocytopenias and thrombocytopenia due to hypersplenism
* Chronic active hepatitis
* Those infected with HIV
* Patients receiving concomitant radiotherapy
* Gravid females
* Congenital thrombocytopenias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population would consist of adult female and male subjects of all ethnic persuasions in good general health apart from thrombocytopenia, bone marrow aplasia, myelodysplasia, or active malignancy requiring therapy. Vulnerable strata of the hospital population will not be recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Increased platelet density | 12 months

SECONDARY OUTCOMES:
mean platelet mass | 12 months

OTHER OUTCOMES:
Platelet mass distribution width | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mala Varma, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Roosevelt Hospital, New York, New York, United States